CLINICAL TRIAL: NCT04848441
Title: Risk of COVID-19 Infection After Vaccination: A Nationwide Study Comparing BNT162b2, mRNA-1273 and ChAdOx1
Brief Title: Risk of COVID-19 Infection After Vaccination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: VACC-COV-19
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Vaccination; Infection; Covid19
Keywords: COVID-19; Vaccination; Nationwide observational study
MeSH Terms: conditions — Infections; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The COVID-19 vaccines BNT162b2, mRNA-1273 and ChAdOx1 — The purpose of the study is to compare the effects of BNT162b2, mRNA-1273 and ChAdOx1 with respect to incident COVID-19 infection of different severities.

SUMMARY:
The purpose of this observational nationwide study is to evaluate the effects of three different COVID-19 vaccines for the outcome of different severities of incident COVID infection.

ELIGIBILITY:
Inclusion Criteria:

* Living in Sweden and vaccinated with BNT162b2, mRNA-1273 or ChAdOx1
* All individuals with a previous COVID-19 infection
* Controls matched 1:1 to the groups above

Exclusion Criteria:

* None

Ages: 0 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will contain all Swedish citizens vaccinated with BNT162b2, mRNA-1273 or ChAdOx1, all Swedish citizens diagnosed with COVID-19, and a control group matched 1:1 on birth year, sex and municipality to the first two groups.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Incident COVID-19 infection | Up to six months after vaccination
  Four different severities: Being diagnosed, hospitalized, ICU-care and death within 30 days of diagnosis

IPD SHARING:
Plan to Share IPD: No